CLINICAL TRIAL: NCT02062528
Title: Evaluation de l'efficacité Des Acides Gras oméga 3 Hautement concentrés en EPA Sur Les bouffées de Chaleur, Chez Des Femmes en période de péri-ménopause et ménopause : étude Monocentrique, en Groupes parallèles, contrôlée, randomisée vs Placebo
Brief Title: Hot Flashes and Omega 3
Acronym: BOOM3
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vivatech (Industry)
Collaborators: Centre d'Investigation Clinique de Grenoble CIC1406 (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DCIC 13 15
Record Dates: First submitted 2014-02-12; First posted 2014-02-13 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Hot Flashes; Fatty Acids; Menopause
Keywords: EPA
MeSH Terms: conditions — Hot Flashes | interventions — Fatty Acids, Omega-3

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega-3 fatty acids (Experimental): 3 capsules each day during 8 weeks
  Interventions: Dietary Supplement: omega-3 fatty acids
- placebo (Placebo Comparator): 3 capsules each day during 8 weeks
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: omega-3 fatty acids — highly dosed in EPA
  Other Names: groupe actif
  Arms: omega-3 fatty acids
Dietary Supplement: placebo
  Arms: placebo

SUMMARY:
The main objective is to evaluate the effects of omega-3 fatty acids on hot flashes frequency.

ELIGIBILITY:
Inclusion Criteria:

* menopause or peri menopause
* complaining of hot flashes
* social security affiliation
* informed consent form signed

Exclusion Criteria:

* primary pathology which can lead to hot flashes
* allergy to omega-3 fatty acids
* allergy to sea products
* High consumption of fat fish or produced by the sea
* iatrogenic hot flashes
* actual omega-3 fatty acids consumption or in the 3 last months.
* consumption of drug or other products for hot flashes in the last month
* protected persons (L1121-5 to L1121-8 of French Public health code)

Min Age: 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2014-03; Primary Completion 2015-05 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
hot flashes frequency | 1 to 8 week
  ANOVA by repeated measures

SECONDARY OUTCOMES:
hot flashes frequency difference | 4 week and 8 week
  difference betwwen week8 and week4 and week0
diurnal hot flashes | week 1 to 8
  ANOVA and difference
night hot flashes | week 1 to 8
  ANOVA and difference
vasomotors disorders | week 1 to week 8
  ANOVA and differences
Pittsburgh Sleep Quality Index (PSQI) | week 0 and week 8
  sleep quality
HFRDIS | week 0 and week 8
  quality of life
The Menopause-Specific Quality of Life (MENQOL) | week 0 and week 8
  quality of life
Weight | week 0 and week 8
fatty acids dosage | week 0 and week 8
  fatty acids dosage
number of adverse events | week 0 to week 8

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Luc CRACOWSKI, MD-PhD, Principal Investigator — Centre d'investigation clinique CIC1406
Locations (1):
- Centre d'investigation clinique CIC1406, Grenoble Cedex9, France